CLINICAL TRIAL: NCT04996615
Title: Peking University People's Hospital Breast Center
Brief Title: Artificial Intelligence Analysis for Magnetic Resonance Imaging in Screening Breast Cancer in High-risk Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Shu Wang, Director of Breast Center, Peking University People's Hospital
Other Study IDs: AI-BMRI
Record Dates: First submitted 2021-07-21; First posted 2021-08-09 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer; Magnetic Resonance Imaging
Keywords: breast cancer; screening; high risk women; magnetic resonance imaging; deep learning
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- high risk population: women at high risk of breast cancer undergoing enhanced MRI
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Use Convolutional Neural Networks Analysis for Classification of Contrast-enhancing Lesions at Multiparametric Breast MRI. Build an abbreviated protocal, and investigate whether an abbreviated protocol was suitable for breast magnetic resonance imaging screening for breast cancer in high-risk Chinese women, which can shorten the examination time and avoid enhanced imaging while ensuring the accuracy of the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing full sequence BMRI examination
* Written informed consent and complete the clinical data questionnaire
* Through the follow-up database, at least 6 months of follow-up results can be obtained to determine whether the diagnosis result is negative/benign/malignant; for patients who need pathological biopsy, the pathological biopsy results shall prevail to determine the lesion benign/malignant.

Exclusion Criteria:

* The breast had received radiotherapy, chemotherapy, biology and other treatments before BMRI.
* Signs or symptoms of breast disease
* There are contraindications for breast-enhanced MRI examinations such as allergy to contrast agents.
* Patients during lactation or pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female
Study Population: 23
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
screening yield | 5 years
  compare the rates of detection of breast cancers in the screening of high-risk populations between the Breast MRI full sequence, contrast-enhanced and non-contrast-enhanced sequence.

SECONDARY OUTCOMES:
The accuracy of radiologists and deep learning models | 5 years
  compare the sensitivity，specificity， positive predictive value and negative predictive value of breast tumor detection by radiologists and deep learning models.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking university people's hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No